CLINICAL TRIAL: NCT04628663
Title: Effects of Systemic Administration of Dexmedetomidine on Intraocular Pressure During Scheduled Spine Surgeries in a Prone Position. Prospective, Randomized, Double-blinded Study.
Brief Title: Effects of Dexmedetomidine on Intraocular Pressure During Scheduled Spine Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Paraskevi Matsota, Prof of Anaesthesiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DEXIOPSPS
Record Dates: First submitted 2020-11-05; First posted 2020-11-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-03

CONDITIONS: Intraocular Pressure
MeSH Terms: interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Placebo -controlled, Double-Blinded clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Not aware of the study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEX group (Active Comparator): Dexmedetomidine given at a bolus dose of 1,0 μg/kg 10min before induction of anesthesia and then after as a continuous infusion 0,4-0,8 μg/kg/h until the end of the surgery.
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): Normal saline given as a bolus dose 10min before induction of anesthesia and then after as a continuous infusion until the end of the surgery.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Administration
  Other Names: Dexmed
  Arms: DEX group
Other: Normal Saline — Administration
  Other Names: Saline
  Arms: Placebo group

SUMMARY:
The aim of this study is to examine the effects of intraoperative systemic use of dexmedetomidine on the intraocular pressure (IOP) in patients undergoing spine surgeries in a prone position under general anesthesia.

DETAILED DESCRIPTION:
The study is a Prospective, Randomized, Placebo -controlled, Double-Blinded clinical trial Adult patients with an ASA physical status of class I, II or III who are scheduled for an elective spine surgery in prone position under general anesthesia will be included in the study.

The patients will be randomized with closed envelope manner into two groups: the group of dexmedetomidine and the group of normal saline.

In the dexmedetomidine group (DEX group), bolus dose 1,0 μg/kg of dexmedetomidine will be administered in 10min before induction to anesthesia and 0,4-0,8 μg/kg/h of dexmedetomidine will be infused continuously until the end of the surgery.

In the saline group (placebo group), the same volume of saline will be administered in an identical way.

All study medication will be prepared by an independent anesthesiologist who is not associated in the study (who will hold the randomization codes until the end of the study).

All patients will receive the same type of anaesthesia (TIVA with propofol) and postoperative analgesia including paracetamol 1gr iv (4 times/day) and continuous wound infiltration with ropivacaine 0.2% 5ml/h for 48 postoperative hours.

Basic monitoring for the study includes:

ECG, Invasive and noninvasive blood pressure, Heart Rate, EtCO2, SpO2, Cardiac Output (CO), Stroke Volume (SV), Stroke Volume Variation (SVV), Patient State index (PSi), IOP, Urine output.

Measurements

The measurement of IOP will be conducted in both eyes with Icare PRO tonometer by an ophthalmologist who will not know in which group the patient is in the below predefined time points:

* T1: before administration of the study drug
* T2: after administration of the bolus dose of the study drug
* T3: after tracheal intubation
* T4: just before prone position
* T5: just after prone position
* T6: 30min after T5
* T7: 60min after T6
* T8: 120min after T7
* T9: 180min after T8
* T10: at the end of the surgery and the patient in supine position At the time of each tonometer reading the following data set is collected: MAP, heart rate, EtCO2, SpO2, CO, SV, SVV, urine output, Psi, IOP. Moreover OPP will be calculated as MAP minus IOP.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing scheduled spine surgery performed in prone position under general anaesthesia

Exclusion Criteria:

* Patients who refuse to be a part of the study
* Patients with previous eye surgery
* Preexisting eye disease (e.g glaucoma)
* Allergy to the study drug or any drug which is in the trial
* Preoperative unstable hemodynamics

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | Up to 15 minutes after the end of operation
  The measurement of IOP will be conducted in both eyes with Icare PRO tonometer by an ophthalmologist at predefined time points

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevi Matsota, Prof, Study Chair — 2nd Department of Anesthesiology, Attikon University Hospital
Locations (1):
- 2nd Department of Anesthesiology, Attikon University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No